CLINICAL TRIAL: NCT02014675
Title: SD01 Registry (SD01 ICD Lead)
Acronym: SD01 Registry
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 67 (TA108)
Record Dates: First submitted 2013-12-04; First posted 2013-12-18 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia; Heart Failure
Keywords: ICD; CRT-D; Lead
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SD01 ICD lead
  Interventions: Device: SD01 ICD lead

INTERVENTIONS:
Device: SD01 ICD lead

SUMMARY:
This registry is designed to gather further evidence, in addition to the SD01 Master Study, for the safety and efficacy of the SD01 ICD lead.

ELIGIBILITY:
Inclusion Criteria:

* Meet a standard indication for ICD/CRT-D therapy
* First ICD/CRT-D implantation or upgrade from pacemaker
* Signed informed consent form
* Willing to participate for the whole duration of the registry
* Patient accepts Home Monitoring concept and is able to activate and use the Cardiomessenger
* Patient has legal capacity and ability to consent

Exclusion Criteria:

* Meet a standard contraindication for an ICD/CRT-D therapy
* Age <18 years
* Pregnant or breast-feeding women
* Cardiac surgery planned within the next six months
* Enrollment in another cardiac clinical investigation with active treatment arm
* Mechanical tricuspid valve prosthesis or severe tricuspid valve disease
* Dexamethasone acetate intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICD/CRT-D (cardiac resynchronization therapy plus defibrillator) indication
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
SADE-free rate | 10 years

OTHER OUTCOMES:
Pacing threshold of SD01 | 3-month follow-up
Sensing amplitude of SD01 | 3-month follow-up
Device deficiencies | 10 years
Long-term pacing impedance, pacing threshold, sensing amplitude and painless shock impedance of SD01 and other leads, if applicable | 10 years
Analysis of arrhythmias and their treatment | until 3-month follow-up
ICD/CRT-D system performance | 10 years
SD01 implantation information, handling and operation time record | Implantation

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - DRK Klinikum Berlin-Köpenick, Berlin
  - Vivantes Humboldt Klinikum Berlin, Berlin
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Klinikum Leverkusen, Leverkusen
  - University Clinic of Schleswig-Holstein, Lübeck
  - Carl-von-Basedow Klinik, Merseburg
  - Marienkrankenhaus Papenburg, Papenburg
  - DRK Krankenhaus Moelln-Ratzeburg, Ratzeburg
  - SRH Zentralklinikum Suhl, Suhl
  - Universitätsklinik Würzburg, Würzburg